CLINICAL TRIAL: NCT02268396
Title: An Open-Label, Multi-Center, Dose Indicator Study of Glycopyrronium and Formoterol Fumarate (GFF) Metered Dose Inhaler (MDI) in Adult Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Glycopyrronium and Formoterol Fumarate (GFF) Metered Dose Inhaler (MDI) Dose Indicator Study in Adults With Moderate to Very Severe COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT003016-00
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (Experimental): Glycopyrronium and Formoterol Fumarate Metered-dose Inhaler (GFF MDI), PT003
  Interventions: Drug: Glycopyrronium and Formoterol Fumarate Metered-dose Inhaler

INTERVENTIONS:
Drug: Glycopyrronium and Formoterol Fumarate Metered-dose Inhaler — GFF MDI administered as 2 inhalations BID
  Other Names: GFF MDI, PT003

SUMMARY:
This is an open-label, multi-center study to evaluate the accuracy, reliability and functionality of the Glycopyrronium and Formoterol Fumarate (GFF) Metered Dose Inhaler (MDI) dose indicator in adult subjects with moderate to very severe COPD over a 4-week Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Give their signed written informed consent to participate.
* Are at least 40 years of age and no older than 80 at Visit 1.
* A female of non-child bearing potential or child bearing potential, has a negative serum pregnancy test, and agrees to approved contraceptive methods.
* COPD Diagnosis: Subjects with an established clinical history of COPD as defined by the American Thoracic Society(ATS)/European Respiratory Society (ERS).
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* FEV1/FVC ratio of <0.70.
* Post-bronchodilator FEV1 must be ≥ 30% and <80% predicted normal value calculated using the Third National Health and Nutrition Examination Survey (NHANES III) reference equations, and must also be greater than or equal to 750 mL.
* Subject is willing and, in the opinion of the Investigator, able to adjust current COPD therapy as required by the protocol.

Exclusion Criteria:

* Pregnancy, nursing females or subjects trying to conceive.
* Clinically significant neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, hematological, psychiatric, or other medical illness that would interfere with participation in this study.
* Current primary diagnosis of asthma.
* History of ECG abnormalities.
* Poorly controlled or worsening COPD prior to Screening or during the Screening Period.
* Clinically significant bladder neck obstruction or urinary retention.
* Male subjects with a trans-urethral resection of prostate (TURP) or full resection of the prostate within 6 months prior to Screening.
* Cancer that has not been in complete remission for at least five years.
* Inadequately treated glaucoma.
* History of allergic reaction or hypersensitivity to any component of the formulations used in this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Director — Pearl Therapeutics
Locations (10):
- United States (10):
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Tampa, Florida
  - Pearl Investigative Site, Winter Park, Florida
  - Pearl Investigative Site, Charlotte, North Carolina
  - Pearl Investigative Site, Columbus, Ohio
  - Pearl Investigative Site, Medford, Oregon
  - Pearl Investigative Site, Greenville, South Carolina
  - Pearl Investigative Site, Rock Hill, South Carolina
  - Pearl Investigative Site, Spartanburg, South Carolina
  - Pearl Investigative Site, Richmond, Virginia

REFERENCES:
- [Derived] Pudi K, Feldman G, Fakih F, Mack P, Maes A, Siddiqui S, St Rose E, Reisner C. An Open-Label Study Evaluating the Performance of the Dose Indicator in a Metered Dose Inhaler Delivering Glycopyrrolate and Formoterol Fumarate in Patients with Moderate-to-Very Severe Chronic Obstructive Pulmonary Disease. J Aerosol Med Pulm Drug Deliv. 2019 Feb;32(1):40-46. doi: 10.1089/jamp.2018.1466. Epub 2018 Nov 1. PMID 30335559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 10 study sites in the United states from November 2014 - January 2015. The entire study period was scheduled to take approximately 6 weeks for each individual subject. The study was anticipated to run for approximately 6 months.
Pre-assignment Details: Study was an open-label, multi center study to evaluate the accuracy, reliability, and functionality of GFF MDI dose indicator in adult subjects with moderate to very severe COPD over a 4-week treatment period.
Groups:
- GFF MDI (PT003): GFF MDI 14.4/9.6 μg
Period: Overall Study
Arm/Group | GFF MDI (PT003)
Started | 138
Completed | 126
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Administrative | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Protocol-Specified Criteria | 2
Not completed — 2 Subjects no Day 29 Assessment | 2

BASELINE CHARACTERISTICS:
Population: 126 received treatment on Day 1 and 29, 10 prematurely discontinued, 2 with no assessment on Day 29.
Arm/Group | GFF MDI (PT003)
Number analyzed (Participants) | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (8.3)
Gender [Count of Participants; unit: Participants]
  Female | 68
  Male | 70

OUTCOME MEASURES:

1. Primary Outcome: Dose Indicator Actuation Consistency: Percentage of Devices in Agreement Between CRF-Based Dose Indicator Actuation Count
Description: Dose Indicator Actuation Consistency: Percentage of Devices in Agreement Between CRF-Based Dose Indicator Actuation Count and Subject-Reported Actuation Count at the Last Available Visit: ITT Population
Time Frame: Over the life of the canister/120 puffs - up to 4 weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | GFF MDI (PT003)
Number analyzed (Participants) | 137
Percentage | 96.4 (18.9) [0 to 130]

2. Secondary Outcome: Percentage of Devices in Agreement Between eCRF-Based Dose Indicator Actuation Count and Weight-Based Actuation Count at the Last Available Visit
Description: Percentage of devices whose number of actuations counted at the end of the study, using the dose indicator reading, was consistent (±20 actuations) with the number of actuations used as estimated by the change in MDI weight
Time Frame: Over the life of the canister/120 puffs - up to 4 weeks
Population: ITT Population
Measure: Number; unit: Percentage of Devices
Arm/Group | GFF MDI (PT003)
Number analyzed (Participants) | 137
Percentage of Devices | 86.9 (19.0) [18 to 130]

3. Secondary Outcome: Percentage of Devices in Agreement Between Laboratory-Advanced Dose Indicator Actuation Count and Subject-Reported Actuation Count at the Last Available Visit
Description: Percentage of devices whose number of actuations counted at the end of the study, using the lab-advanced dose indicator reading, was consistent (±20 actuations) with the number of actuations used as reported by the subject
Time Frame: Over the life of the canister/120 puffs - up to 4 weeks
Population: ITT Population
Measure: Number; unit: Percentage of devices
Arm/Group | GFF MDI (PT003)
Number analyzed (Participants) | 132
Percentage of devices | 96.2 (19.0) [0 to 130]

4. Secondary Outcome: Percentage of Devices in Agreement Between Laboratory-advanced Does Indicator Actuation and Weight-based Actuation Count at Last Available Visit.
Description: as for outcome 2
Time Frame: Over the life of the canister/120 puffs - up to 4 weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | GFF MDI (PT003)
Number analyzed (Participants) | 132
Percentage | 75.0 (19.0) [17 to 171]

5. Secondary Outcome: Percentage of Devices Where the Dose Indicator Actuation Count is >20 Less Than the Subject-reported Actuation Count (Undercount)
Description: Percentage of devices where the dose indicator actuation count is >20 less than the subject-reported actuation count (undercount)
Time Frame: Over the life of the canister/120 puffs - up to 4 weeks
Population: ITT Population
Measure: Number; unit: Percentage
Arm/Group | GFF MDI (PT003)
Number analyzed (Participants) | 132
Percentage | 2.9 (2.9) [17 to 171]

6. Secondary Outcome: Percentage of Correct Advances (±2 or ±4 Actuations) of the Dose Indicator Based on Subject-reported Actuation Count
Description: Percentage of Correct Advances (±2 or ±4 Actuations) of the Dose Indicator Based on Subject-reported Actuation Count
Time Frame: Over the life of the canister/120 puffs - up to 4 weeks
Population: ITT Population
Measure: Number; unit: Percentage of correct advances
Arm/Group | GFF MDI (PT003)
Number analyzed (Participants) | 132
Percentage of correct advances
  Correct within ±2 actuations | 87.3 [17 to 171]
  Correct within ±4 actuations | 93.2

ADVERSE EVENTS:
Time Frame: AEs occurring between when signed consent and randomized reported as SAEs up to 14 days following last dose of study drug. AEs occurring at time of and following first study drug administration were reported and followed until stabilized/resolved.
Description: Safety population included all participants who received at least one dose of investigational drug and had safety data available (Note: A subject who used the GFF MDI, but took less than 1 full dose of treatment qualified for this population.)
Arm/Group | GFF MDI (PT003)
Serious Adverse Events (participants affected / at risk) | 3/138
Other Adverse Events (participants affected / at risk) | 10/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (PT003) (N=138)
COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Chronic Obstructive pulmonary disease
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (PT003) (N=138)
COPD (Respiratory, thoracic and mediastinal disorders) | 10 (11) — Chronic Obstructive Pulmonary disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.